CLINICAL TRIAL: NCT05427851
Title: Effect Of Diode Laser And Platelet Rich Fibrin In Regenerative Pulpotomy Of Mature Permanent Molars With Irreversible Pulpitis (A Randomized Controlled Clinical Trial)
Brief Title: Diode Laser Pulpotomy of Mature Permanent Molars With Irreversible Pulpitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Darinemamdouh
Record Dates: First submitted 2022-06-12; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Irreversible Pulpitis
MeSH Terms: interventions — Pulpotomy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Group I: Platelet rich Fibrin (PRF) and Biodentine (Experimental)
  Interventions: Procedure: pulpotomy
- Group II: Diode Laser and Biodentine (Experimental)
  Interventions: Procedure: pulpotomy; Device: Diode laser - fonalaser
- Group III: Diode laser + PRF + Biodentine (Experimental)
  Interventions: Procedure: pulpotomy; Device: Diode laser - fonalaser

INTERVENTIONS:
Procedure: pulpotomy — coronal pulp tissue removal followed by radicular pulp hemostasis them applying a pulp capping material
Device: Diode laser - fonalaser — diode laser beam application
  Arms: Group II: Diode Laser and Biodentine; Group III: Diode laser + PRF + Biodentine

SUMMARY:
Thirty six patients are included in this study. For each patient, a pulpotomy procedure is performed.

DETAILED DESCRIPTION:
For each patient, a pulpotomy procedure is done. Group I (n=12) pulpotomy is performed and hemostasis is achieved by applying NaOCl, then the radicular pulp is covered with Platelet Rich Fibrin (PRF) and capped with Biodentine, Group II (n=12) pulpotomy is done as in group I and hemostasis is achieved using diode laser and remaining pulp is capped with Biodentine, Group III (n=12) pulpotomy is performed and hemostasis is achieved as in group II then radicular pulp is covered with PRF then capped with Biodentine, The teeth are then restored with Glass ionomer cement followed by composite restoration. Pain is recorded every 24 hours for 7 days after intervention. Clinical and radiographic follow-up are done at 1,3,6,9 and 12 months. Cone beam computed tomography (CBCT) is done immediate postoperative and will be used for the assessment of the outcome of the pulpotomy procedure at the end of the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18 and 40 years of age.
2. Deep caries in a permanent lower molar with mature roots.
3. Clinical diagnosis of symptomatic irreversible pulpitis
4. No signs of pulpal necrosis including sinus tract or swelling.
5. Vital bleeding pulp tissue should be present in all canals after complete pulpotomy.
6. The tooth is restorable.

Exclusion Criteria:

1. Patients with systemic disease.
2. Negative response to cold testing.
3. Presence of sinus tract or swelling.
4. No pulp exposure after caries excavation.
5. Bleeding could not be controlled
6. Absence of bleeding from any of the canals.
7. Teeth with radiographic signs of internal resorption.
8. Pulpal calcifications.
9. Non-restorable teeth

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
regenerative pulpotomy success | 12 months
  Assessing the clinical and radiographic success rate of the regenerative pulpotomy. • Teeth were considered as clinical success if patients had lack of pain (spontaneous or on chewing), sinus tract or swelling, pathological mobility, and had intact coronal restoration.( procedure done in permanent mature teeth with irreversible pulpitis.
  Treatment was considered radiographically successful if no pathosis was evident on the recall radiograph such as root resorption, no furcal or periapical rarefaction. Periapical Index (PAI) was used to evaluate the periapical tissue condition by comparing the pre-operative radiographs with the follow-up radiographs.

SECONDARY OUTCOMES:
Postoperative pain | 7 days
  To evaluate the effect of Diode laser on decreasing the immediate postoperative pain. Postoperative pain was recorded on Numerical Rating Pain Scale (NRS) that was given to the patient in Arabic language to record his pain experience every 24 hours until the seventh day after the first appointment.
  Pain on the NRS was further categorized as:(0)no pain, (1-3) mild, (4-6) moderate, (7-10) Severe pain.

OTHER OUTCOMES:
Dentine bridge formation | 12 months
  To evaluate the effect of Diode laser on the enhancement of dentin bridge formation following pulpotomy procedure using CBCT.

CONTACTS AND LOCATIONS:
Overall Officials: Raef A sherif, PhD, Study Director — Professor of Endodontics, Faculty of Dentistry, Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt